CLINICAL TRIAL: NCT04112004
Title: Effect of Perioperative Delta Sodium on Outcomes in Liver Transplant Recipients
Brief Title: Effect Of Delta Sodium on the Postoperative Outcomes in Liver Transplant Recipients
Acronym: SOLT
Status: Completed | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Principal Investigator, Karthik Ponnappan T, Consultant, Institute of Liver and Biliary Sciences, India
Other Study IDs: ILBS - Liver Transplant-1
Record Dates: First submitted 2019-06-30; First posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Liver Transplant; Complications; Perioperative/Postoperative Complications; Electrolyte Disturbance
Keywords: liver transplantation; perioperative sodium; sodium
MeSH Terms: conditions — Postoperative Complications | interventions — Outcome Assessment, Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver Transplant Recipients: All elective liver transplant recipients done between study period
  Interventions: Other: Collecting sodium reports and outcome measures

INTERVENTIONS:
Other: Collecting sodium reports and outcome measures

SUMMARY:
We analyzed the association of delta sodium levels with their effect on post liver transplant outcomes in consecutive patients undergoing liver transplantation. Records were analyzed for electrolytes and outcome measures, and data was analyzed.

DETAILED DESCRIPTION:
Preoperative hyponatremia was identified in patients. The mean change in sodium in hyponatremic patients was compared with inpatients with normal sodium levels. The impact of the delta sodium levels with short-term outcomes, such as duration of intubation, intensive care unit length of stay were analyzed with univariate and multivariate logistic regression analyses.

ELIGIBILITY:
Inclusion Criteria:

* All liver transplant recipients between Jan 2011 to Jan 2017
* Records available

Exclusion Criteria:

* Acute fulminant liver failure
* All patients less than 18 years
* Re operated cases
* Pregnant patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver transplant recipients more than 18 years in ILBS during study period
Sampling Method: Non-Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
change in serum sodium in liver transplant recipients | 1 day
  difference between baseline and postoperative sodium in liver transplant recipients
post transplant mortality | 1 month
  post transplant mortality after liver transplantation

SECONDARY OUTCOMES:
post operative neurological complications | 1 month
  Post operative neurological complications after liver transplantation
duration of mechanical ventilation | 1 month
  duration of mechanical ventilation after liver transplantation
Duration of hospital stay | 1 month
  Hospital stay after liver transplantation
Duration of ICU stay | 1 month
  Duration of ICU stay after liver transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Karthik T Ponnappan, DM, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT04112004/Prot_SAP_000.pdf